CLINICAL TRIAL: NCT05962684
Title: A Greek-designed Enhanced Recovery After Surgery (ERAS) Protocol in Elective Cranial Neurosurgical Procedures: An Observational Study
Brief Title: A Greek-designed ERAS Protocol in Elective Craniotomy
Acronym: ERAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor in Anesthesiology, University of Thessaly
Other Study IDs: ERAS Craniotomy
Record Dates: First submitted 2023-07-12; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: ERAS; Craniotomy
Keywords: ERAS; Craniotomy; Perioperative management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERAS
  Interventions: Other: ERAS

INTERVENTIONS:
Other: ERAS — Implementation of ERAS protocol in elective craniotomy patients

SUMMARY:
The implementation of ERAS protocol in elective cranial neurosurgical cases in a tertiary hospital.

DETAILED DESCRIPTION:
In this study, the investigators have integrated the most current data from literature aiming to investigate the effectiveness of a contemporary ERAS protocol for elective cranial neurosurgical cases in a tertiary hospital. The hypothesis is that the implementation of such protocol will shorten the postoperative length of stay, minimize the complication rates, and improve the overall clinical status of patients undergoing elective craniotomy compared to the standard perioperative care

ELIGIBILITY:
Inclusion Criteria:

* Medically suitable for elective craniotomy
* ASA-PS I-III

Exclusion Criteria:

* traumatic lesions
* pathology requiring emergent surgery
* preoperative loss of consciousness
* severe co-morbidities that may affect postoperative recovery (e.g. paralysis, autoimmune diseases, myocardial or severe infarction, heart, liver or lung malfunction, severe mental illness etc.)
* recurrent tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective craniotomy
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Length of Stay | up to 7 days
  The days the patient stays in hospital

SECONDARY OUTCOMES:
Pain score | Postoperative Day 1 to discharge, an average of 7 days
  Pain intensity as measured by Visual Analogue Scale (VAS)
Mental status | 1 day at discharge
  Mental status as measured by Glasgow Coma Scale (GCS) Minimum value : 3 Maximum value : 15 Higher scores mean a better outcome
Patient's satisfaction | 1 day at discharge and 1 month postoperatively
  Patient's satisfaction as measured by a Likert Scale
Anxiety and Depression | Preoperatively, second postoperative day and one month postoperatively
  Anxiety and Depression level as measured by Hospital Anxiety and Depression Scale (HADS)
Personality Index | Preoperatively, second postoperative day and one month postoperatively
  Personality Index as measured by TIPI

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutolglou, MD, PhD, Study Director — University of Thessaly; Konstantinos Fountas, MD, PhD, Study Chair — University of Thessaly
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang L, Cai H, Wang Y, Liu J, Chen T, Liu J, Huang J, Guo Q, Zou W. Enhanced recovery after elective craniotomy: A randomized controlled trial. J Clin Anesth. 2022 Feb;76:110575. doi: 10.1016/j.jclinane.2021.110575. Epub 2021 Nov 2. PMID 34739947
- [Result] Wang Y, Xue YF, Zhao BF, Guo SC, Ji PG, Liu JH, Wang N, Chen F, Zhai YL, Wang Y, Xue YR, Gao GD, Qu Y, Wang L. Real-World Implementation of Neurosurgical Enhanced Recovery After Surgery Protocol for Gliomas in Patients Undergoing Elective Craniotomy. Front Oncol. 2022 May 24;12:860257. doi: 10.3389/fonc.2022.860257. eCollection 2022. PMID 35686112
- [Result] Elayat A, Jena SS, Nayak S, Sahu RN, Tripathy S. "Enhanced recovery after surgery - ERAS in elective craniotomies-a non-randomized controlled trial". BMC Neurol. 2021 Mar 19;21(1):127. doi: 10.1186/s12883-021-02150-7. PMID 33740911
- [Result] Wang Y, Liu B, Zhao T, Zhao B, Yu D, Jiang X, Ye L, Zhao L, Lv W, Zhang Y, Zheng T, Xue Y, Chen L, Sankey E, Chen L, Wu Y, Li M, Ma L, Li Z, Li R, Li J, Yan J, Wang S, Zhao H, Sun X, Gao G, Qu Y, He S. Safety and efficacy of a novel neurosurgical enhanced recovery after surgery protocol for elective craniotomy: a prospective randomized controlled trial. J Neurosurg. 2018 Jun 22;130(5):1680-1691. doi: 10.3171/2018.1.JNS171552. Print 2019 May 1. PMID 29932379
- [Result] Stumpo V, Staartjes VE, Quddusi A, Corniola MV, Tessitore E, Schroder ML, Anderer EG, Stienen MN, Serra C, Regli L. Enhanced Recovery After Surgery strategies for elective craniotomy: a systematic review. J Neurosurg. 2021 May 7;135(6):1857-1881. doi: 10.3171/2020.10.JNS203160. Print 2021 Dec 1. PMID 33962374
- [Result] Agarwal P, Frid I, Singer J, Zalatimo O, Schirmer CM, Kimmell KT, Agarwal N. Neurosurgery perception of Enhanced Recovery After Surgery (ERAS) protocols. J Clin Neurosci. 2021 Oct;92:110-114. doi: 10.1016/j.jocn.2021.07.044. Epub 2021 Aug 7. PMID 34509236